CLINICAL TRIAL: NCT01542255
Title: Metronomic Therapy in Patients With Metastatic Melanoma: A Phase II Study of Low Dose Vinblastine, Cyclophosphamide, and Dacarbazine
Brief Title: Metronomic Therapy in Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual not allowing to support statistical endpoints
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1010; 22362 (Other: Committee for the Protection of Human Subjects)
Record Dates: First submitted 2012-01-17; First posted 2012-03-02 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2014-09

CONDITIONS: Metastatic Melanoma
Keywords: Metronomic Therapy; Metastatic Melanoma; Vinblastine; Cyclophosphamide; Dacarbazine
MeSH Terms: conditions — Melanoma | interventions — Vinblastine; Cyclophosphamide; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined Low Dose Treatment (Experimental): A cycle of therapy is 3 weeks of continuous dosing with a 1 week rest.
  Schema of treatment is:
  1 mg/m2 vinblastine three times a week iv 60 mg/m2 cyclophosphamide by mouth 15 mg/m2 dacarbazine three times a week iv
  Interventions: Drug: vinblastine; Drug: Cyclophosphamide; Drug: dacarbazine

INTERVENTIONS:
Drug: vinblastine — 1 mg/m2 vinblastine given three times per week administered intravenously.
  Other Names: Velban
Drug: Cyclophosphamide — 60 mg/m2 cyclophosphamide taken orally every day for 3 weeks with one week rest
  Other Names: Cytoxan
Drug: dacarbazine — 15 mg/m2 dacarbazine given three times per week for 3 weeks with 1 week rest
  Other Names: DTIC

SUMMARY:
SUMMARY: Metronomic Therapy in Patients with Metastatic Melanoma: A Phase II Study of Low Dose Vinblastine, Cyclophosphamide, and Dacarbazine.

Patients with measurable metastatic melanoma are eligible. All patients will be treated as outlined below with combined vinblastine, cyclophosphamide, and dacarbazine. Patients will be treated continuously, until evidence of progression of disease, or for up to two cycles following disappearance of all disease. A cycle will be defined as three weeks of continuous therapy with a one week rest.

DETAILED DESCRIPTION:
Low dose continuous chemotherapy, called metronomic chemotherapy, is designed to target vascular cells and inhibit tumor growth and metastasises. A recent study in a melanoma mouse model has identified low dose vinblastine, cyclophosphamide and dacarbazine as a treatment which improves the animal's survival and is superior to full dose dacarbazine alone. This clinical trial seeks to translate this laboratory model directly into metastatic melanoma patients.

ELIGIBILITY:
* Metastatic melanoma with measurable disease
* Patients must be at least 4 weeks from their last immunotherapy, radiation, surgery or chemotherapy (6 weeks for nitrosoureas) and recovered from all ill
* Karnofsky Performance Status ≥60%
* Life expectancy ≥ twelve weeks
* Adequate end organ function
* Women should not be lactating and, if of childbearing age, have a negative pregnancy test within two weeks of entry to the study.
* Appropriate Contraception in both sexes
* The patient must be competent and signed informed consent.

EXCLUSION CRITERIA

* Concomitant second malignancy except for non-melanoma skin cancer, and non-invasive cancer such as cervical CIS, superficial bladder cancer without local recurrence, breast CIS.
* In patients with a prior history of invasive malignancy, less than five years in complete remission.
* Have evidence of significant co-morbid illness such as uncontrolled diabetes - Uncontrolled brain metastasis: Patients with brain metastasis most have been treated with brain radiation therapy or surgery and remain clinically stable for a minimum of 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc S. Ernstoff, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled from 6/2010 to 11/2012 at Dartmouth Hitichcock
Groups:
- Combined Low Dose Treatment: A cycle of therapy is 3 weeks of continuous dosing with a 1 week rest.
  Schema of treatment is:
  1 mg/m2 vinblastine three times a week iv 60 mg/m2 cyclophosphamide by mouth 15 mg/m2 dacarbazine three times a week iv
  vinblastine: 1 mg/m2 vinblastine given three times per week administered intravenously.
  Cyclophosphamide: 60 mg/m2 cyclophosphamide taken orally every day for 3 weeks with one week rest
  dacarbazine: 15 mg/m2 dacarbazine given three times per week for 3 weeks with 1 week rest
Period: Overall Study
Arm/Group | Combined Low Dose Treatment
Started | 7
Analyzed for Time to Progression | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: patients with metastatic melanoma
Arm/Group | Combined Low Dose Treatment
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 65 [48 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Tumor evaluation will be performed every 8 weeks from day 1 of cycle 1 (+/- 1 week) while on therapy assessed by RECIST 1.0 criteria.
Time Frame: From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Measure: Median (Full Range); unit: weeks
Arm/Group | Single Arm
Number analyzed (Participants) | 7
weeks | 3 [3 to 15]

2. Secondary Outcome: Clinical Response Rate
Description: To be assigned a status of partial response or complete response, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 4 weeks after the criteria for response are first met. In the case of stable disease, follow-up measurements must have met the stable disease criteria at least once after study entry at a minimum interval (in general, not less than 6-8 weeks) that is defined in the study protocol
Time Frame: Tumor evaluation will be performed every 8 weeks from day1 of cycle 1 (+ 1 week) while on therapy, clinical response will be assessed no less than 4 weeks after response criteria met.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Low Dose Treatment
Number analyzed (Participants) | 7
Participants
  Stable Disease | 2
  Progressive Disease | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from the time of start of treatment until 30 days after the last dose of treatment. As this study ended prematurely, adverse events were collected only for the seven subjects enrolled over a period of 1 year.
Groups:
- Single Arm: all patients received cyclophosphamide, DTIC and vinblastine
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=7)
alanine aminotransferase increased (Investigations) | 1 (4)
alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2)
Creatinine increased (Investigations) | 3 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema - limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain - extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (7)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
terminated early due to difficulty with scheduling three times per week office treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No